CLINICAL TRIAL: NCT05384210
Title: Effect of Milnacipran Versus Gabapentin or Combination of Both in Fibromyalgia Syndrome
Brief Title: Effect of Milnacipran / Gabapentin in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MFM-IRB، MD.21.12.577
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Milnacipran (Active Comparator): Patients will receive Milnacipran as a mono-therapy will be administered in increment doses for 3 months
  Interventions: Drug: Milnacipran
- Gabapentin (Active Comparator): patients will receive Gabapentin as a mono-therapy will be administered in increment doses for 3 months
  Interventions: Drug: Gabapentin
- Combined gabapentin/milnacipran (Active Comparator): Patients will receive combined gabapentin and milnacipran as a combination therapy will be administered in increment doses for 3 months
  Interventions: Drug: Combined gabapentin/milnacipran

INTERVENTIONS:
Drug: Milnacipran — Milnacipran will be administered according to the treatment recommendations for fibromyalgia, starting with 50 mg once daily for 1 week then increasing to reach 100 mg daily (50 mg twice daily) based on efficacy and tolerability for 3 months.
  Arms: Milnacipran
Drug: Gabapentin — Patients will receive gabapentin (1200 mg twice daily) as a monotherapy. Gabapentin will be administered according to the treatment recommendations for FM patients starting with 400 mg 3 times per day, then increasing the dose to 800 mg 3 times per day with a maximum dose of 2400 mg per day according to efficacy and tolerability for 3 months
  Arms: Gabapentin
Drug: Combined gabapentin/milnacipran — Patients will receive combined gabapentin as group B and MLN as group A
  Arms: Combined gabapentin/milnacipran

SUMMARY:
Gabapentin and milnacipran (MLN) show strong evidence of reduced pain, increased sleep, and improvement in the quality of life in fibromyalgia (FM) patients.

Most FM trials focus primarily on pain reduction with monotherapy. Polypharmacy is commonly used, but supportive evidence is limited.

The gabapentin-MLN combined therapy may be more effective in female patients with FM than their monotherapy.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the analgesic efficacy of gabapentin-MLN as combined or monotherapy on patients with FM.

ELIGIBILITY:
Inclusion Criteria:

* There are no other criteria rather than age and sex

Exclusion Criteria:

* Patient refusal.
* Pregnancy or breastfeeding.
* Active liver disease
* Renal impairment (creatinine clearance < 60 mL/min).
* Documented autoimmune disease.
* Severe chronic obstructive pulmonary disease.
* Recent arrhythmia
* Myocardial infarction
* Stroke.
* Uncontrolled hypertension.
* Glaucoma.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) for pain | 3 months
  Assesses the overall pain of fibromyalgia on a 10 cm pain scale with 0 indicating no pain and 10 indicating the worst pain ever

SECONDARY OUTCOMES:
The Fibromyalgia Impact Questionnaire (FIQ). | 3 months
  Assesses the overall functional ability and the impact of fibromyalgia on the patient's life, with a range from 0-100, 0 indicating no functional impairment or effect of the disease on the patient's life and 100 indicating a very bad and tremendous effect of fibromyalgia on the patient's life.
Leeds Sleep Evaluation Questionnaire | 3 months
  The four aspects of sleep around which the questionnaire is devised (Getting to sleep, GTS; Quality of sleep, QOS; Awakening from sleep, AFS; Behaviour following wakefulness, BFW), and assessing the effect of medication on the quality of sleep each question is a 100 mm line that the patient marks, 0 meaning very bad effect or worsening in sleep pattern, 50 meaning no improvement what so ever with no deterioration and 100 meaning excellent improvement in the sleep pattern

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassin, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Eiad A Ramzy, md, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes, Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completing the study and being accepted for publication.
Access Criteria: The data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients.